CLINICAL TRIAL: NCT03525743
Title: Non-invasive Cardiac Output Monitoring (NICOM) in Critically Ill Patient Undergoing Endotracheal Intubation in ICU
Brief Title: Cardiac Output Monitoring in Critically Ill Patient Undergoing Intubation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nathan J. Smischney, Principal Investigator, Mayo Clinic
Other Study IDs: 16-006354
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Hypotension
Keywords: Intubation
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing intubation: Adhesive gel pads will be placed on patient to measure continuous cardiac output and to calculate stroke volume variation. Other physiologic data will be analyzed in real time using the NICOM (Non invasive cardiac output monitor) device.
  Interventions: Device: NICOM (Non invasive cardiac output monitor)

INTERVENTIONS:
Device: NICOM (Non invasive cardiac output monitor) — Non invasive hemodynamic device utilizing bioreactance

SUMMARY:
Collect hemodynamic data, such as heart rate, blood pressure, and cardiac output to help understand the effect of pre and post intubation.

DETAILED DESCRIPTION:
A Non-invasive physiologic monitor, Non-Invasive Cardiac Output Monitor (NICOM), will be utilized for this study. This is the first completely non-invasive hemodynamic device approved by the FDA and available for clinical use produced by Cheetah Medical and utilizes Bioreactance (Tel Aviv, Israel). It performs accurately and with precision in all patient's studied and requires only 4 adhesive gel pads on the skin to measure continuous cardiac output and to calculate Stroke Volume Variation (SVV). Other physiologic data (blood pressure, total peripheral resistance (TPR), stroke volume (SV), and heart rate) will be analyzed in real time and recorded on the device and downloaded into an excel database. The data on the device will be downloaded weekly onto the excel database and deleted on the device. The Study personnel will be trained in its use prior to study initiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring endotracheal intubation in the intensive care unit.

Exclusion Criteria:

* Patients previously enrolled in this study.
* Patients requiring intubation outside of the intensive care unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Change in cardiac output in critically ill patients undergoing endotracheal intubation | 10 minutes pre intubation,10 minutes post intubation
  change in cardiac output as measured in liters/minute

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Smischney, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - New York University Tisch Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Green RS, Turgeon AF, McIntyre LA, Fox-Robichaud AE, Fergusson DA, Doucette S, Butler MB, Erdogan M; Canadian Critical Care Trials Group (CCCTG). Postintubation hypotension in intensive care unit patients: A multicenter cohort study. J Crit Care. 2015 Oct;30(5):1055-60. doi: 10.1016/j.jcrc.2015.06.007. Epub 2015 Jun 16. PMID 26117220
- [Background] Green R, Hutton B, Lorette J, Bleskie D, McIntyre L, Fergusson D. Incidence of postintubation hemodynamic instability associated with emergent intubations performed outside the operating room: a systematic review. CJEM. 2014 Jan;16(1):69-79. doi: 10.2310/8000.2013.131004. PMID 24424005
- [Background] Smischney NJ, Demirci O, Diedrich DA, Barbara DW, Sandefur BJ, Trivedi S, McGarry S, Kashyap R. Incidence of and Risk Factors For Post-Intubation Hypotension in the Critically Ill. Med Sci Monit. 2016 Feb 2;22:346-55. doi: 10.12659/msm.895919. PMID 26831818
- [Background] Smischney NJ, Beach ML, Loftus RW, Dodds TM, Koff MD. Ketamine/propofol admixture (ketofol) is associated with improved hemodynamics as an induction agent: a randomized, controlled trial. J Trauma Acute Care Surg. 2012 Jul;73(1):94-101. doi: 10.1097/TA.0b013e318250cdb8. PMID 22743378
- [Derived] Smischney NJ, Stoltenberg AD, Schroeder DR, DeAngelis JL, Kaufman DA. Noninvasive Cardiac Output Monitoring (NICOM) in the Critically Ill Patient Undergoing Endotracheal Intubation: A Prospective Observational Study. J Intensive Care Med. 2023 Dec;38(12):1108-1120. doi: 10.1177/08850666231183401. Epub 2023 Jun 15. PMID 37322892
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials